CLINICAL TRIAL: NCT01344122
Title: Medication-Assisted Treatment Implementation in Community Correctional Environments (MATICCE)
Acronym: MATICCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Arizona State University (Other); Friends Research Institute, Inc. (Other); National Development and Research Institutes, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH); Temple University (Other); Texas Christian University (Other); University of California, Los Angeles (Other); University of Connecticut (Other); University of Delaware (Other); University of Kentucky (Other); University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Peter D. Friedmann, Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CJDATS2-001; U01DA016191 (NIH)
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Opioid-Related Disorders; Alcohol-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Alcohol-Related Disorders

ARMS (2):
- KPI training only (Active Comparator): Study sites randomized to this arm will receive a knowledge, perceptions and information (KPI) training for community correctional and treatment staff to address knowledge, perceptions, and information regarding local resources about MAT.
  Interventions: Other: KPI training only
- KPI plus OLI (Experimental): Study sites randomized to this arm will receive the KPI training plus a Organizational Linkage Intervention (OLI) that will: (a) establish a local Pharmacotherapy Exchange Council (PEC) among agencies important for the implementation of MAT in community corrections; (b) facilitate a strategic planning process within the PEC to increase the availability of MAT for opiate and/or alcohol dependent individuals who are on probation/parole; and (c) identify a community corrections coordinator in one of the local agencies to operationalize and implement the strategic plan.
  Interventions: Other: KPI plus OLI

INTERVENTIONS:
Other: KPI training only — See comparison arm description.
  Arms: KPI training only
Other: KPI plus OLI — See experimental arm description.
  Arms: KPI plus OLI

SUMMARY:
The goal of this study is to see whether or not a strategic planning process is able to introduce and sustain improvements in the working relationship between probation/parole departments and community-based addiction treatment agencies that provide medication assisted therapy (MAT) for individuals with opioid or alcohol dependence. In addition, this study seeks to improve probation/parole agency personnel's knowledge and perceptions about MAT, and increase the number of appropriate referrals to community treatment agencies that provide MAT. There are three phases to this study. Phase 1 includes a pilot study to determine the quality and availability of client level records and the collection of baseline data (the pilot study protocol was previously submitted to TMH IRB). Phase 2 will consist of a Knowledge, Perceptions and Information (KPI) intervention during which probation/parole agencies will undergo training to increase knowledge about the effectiveness of MAT, and complete a post training assessment to evaluate the effectiveness of the KPI intervention. During Phase 3, probation/parole agencies will be randomly assigned to a 12-month Organizational Linkage Intervention (OLI) condition or to control (no further intervention). Agencies assigned to the OLI will establish a Pharmacotherapy Exchange Council (PEC) that consists of staff from both the probation/parole and community treatment agencies. The PEC will undergo a strategic planning process to increase the availability of MAT for opiate and/or alcohol dependent individuals who are on probation/parole.

ELIGIBILITY:
Probation/parole or community treatment agency staff.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Opinions About MAT | 6-month follow-up
  Measures knowledge, perceptions, and intentions regarding the use of pharmacotherapy for the treatment of opioid and alcohol dependence. Will be assessed at baseline, post-training, post intervention, and 6-month follow-up.

SECONDARY OUTCOMES:
Interorganizational Relationships | 6-month follow-up
  Will be assessed at baseline, and post intervention (6-month follow-up).
Referrals to Medication Assisted Treatment (MAT) | 6-Month Follow-up
  Estimated numbers of alcohol- and opiate-dependent offenders on Probation/Parole

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD, MPH, Principal Investigator — Rhode Island Hospital

REFERENCES:
- [Derived] Friedmann PD, Wilson D, Knudsen HK, Ducharme LJ, Welsh WN, Frisman L, Knight K, Lin HJ, James A, Albizu-Garcia CE, Pankow J, Hall EA, Urbine TF, Abdel-Salam S, Duvall JL, Vocci FJ. Effect of an organizational linkage intervention on staff perceptions of medication-assisted treatment and referral intentions in community corrections. J Subst Abuse Treat. 2015 Mar;50:50-8. doi: 10.1016/j.jsat.2014.10.001. Epub 2014 Oct 14. PMID 25456091